CLINICAL TRIAL: NCT04974398
Title: A Randomized, Double-blind, Multi-center Phase III Study of Penpulimab (AK105) Combined With Chemotherapy Versus Placebo Combined With Chemotherapy in the First-line Treatment of Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: A Study of Penpulimab (AK105) in the First-line Treatment of Recurrent or Metastatic Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK105-304
Record Dates: First submitted 2021-07-13; First posted 2021-07-23 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — penpulimab; Cisplatin; Carboplatin; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A (study group): Penpulimab plus cisplatin/carboplatin and gemcitabine
  Interventions: Drug: Penpulimab
- Group B (Placebo Comparator): Group B (control group): Placebo plus cisplatin/carboplatin and gemcitabine
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Penpulimab — Arm A: Penpulimab (200 mg, administered on Day 1 of each cycle, Q3W) +cisplatin (80 mg/m2) or carboplatin (AUC 5) (administered on Day 1 of each cycle, Q3W, up to 6 cycles) + gemcitabine (1000 mg/ m2, administered on Days 1 and 8 of each cycle, Q3W, up to 6 cycles), 3 weeks (21 days) per cycle; followed by penpulimab (200 mg, administered on Day 1 of each cycle, Q3W) as maintenance treatment.
  Other Names: cisplatin/carboplatin; gemcitabine
  Arms: Group A
Drug: placebo — Arm B: Placebo (200 mg, administered on Day 1 of each cycle, Q3W) + cisplatin (80 mg/m2) or carboplatin (AUC 5) (administered on Day 1 of each cycle, Q3W, up to 6 cycles) + gemcitabine (1000 mg/m2, administered on Days 1 and 8 of each cycle, Q3W, up to 6 cycles), every 3 weeks (21 days) per cycle; followed by placebo(200 mg, administered on Day 1 of each cycle, Q3W) as maintenance treatment. Subjects in Arm B will have the opportunity to crossover to openlabel treatment with penpulimab monotherapy after radiographic disease progression.
  Other Names: cisplatin/carboplatin; gemcitabine
  Arms: Group B

SUMMARY:
This study is a randomized, double-blind, multi-center phase III clinical study to compare the efficacy and safety of penpulimab combined with chemotherapy and placebo combined with chemotherapy in the first-line treatment of recurrent or metastatic nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed written Informed Consent Form(ICF).
* Main study: Age of ≥ 18 years and ≤ 75 years at the time of enrollment.
* Substudy: Age of ≥ 12 years and < 18 years. Weight≥ 35KG.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Expected survival of ≥ 3 months.
* Histologically or cytologically confirmed nasopharyngeal carcinoma.
* Subjects with primary metastatic (nasopharyngeal carcinoma, stage IVB defined by the Union for International Cancer Control and the American Joint Committee on Cancer Staging System edition 8) nasopharyngeal carcinoma who are not suitable for local treatment or radical treatment; subjects who have a local-regional recurrence and/or distant metastasis more than 6 months after the completion of prior radical treatment (radiotherapy with induction, concurrent, adjuvant chemotherapy)； No systemic treatment has been received for recurrent or metastatic diseases, not amendable to local treatment or have received local treatment for the local-regional recurrent disease
* At least one measurable lesion according to RECIST v1.1;
* Has adequate organ function.
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 150 days after the last dose of study treatment.

Exclusion Criteria:

* Subjects with pathologically diagnosed nasopharyngeal adenocarcinoma or sarcoma.
* Subjects have had another malignancy within 3 years before the first dose, except nasopharyngeal carcinoma. Subjects with other malignancies that have been cured by local therapy such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervix or breast carcinoma in situ are not excluded.
* Participation in treatment with an investigational drug or use of an investigational device within 4 weeks before first study dosing.
* Have previously received immunotherapy, including immune checkpoint inhibitors, immune checkpoint agonists , immune cell therapy, and other treatments against tumor immune mechanism.
* Active autoimmune disease requiring systemic treatment within 2 years prior to initial administration, or as an autoimmune disease that can recur or for which treatment is planned determined by the investigator.
* Active or past history of definite inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis).
* History of immunodeficiency; those who test positive for HIV antibody; current chronic use of systemic corticosteroids or immunosuppressive agents.
* Known active tuberculosis (TB) (suspected of having active TB need to undergo clinical examination for exclusion of such possibility); known active syphilis infection.
* Known history of allotransplantation and allogeneic hematopoietic stem cell transplantation.
* Has known active Hepatitis B or Hepatitis C.
* Active or untreated CNS metastases.
* Subjects with peripheral neuropathy.
* Unresolved toxicity from prior anti-tumor therapy, defined as toxicity that has not recovered .
* Received a live vaccine within 30 days before the first dose or planned to receive a live vaccine during the study.
* Known allergy to any study drug component; known history of serious hypersensitivity to other monoclonal antibodies.
* Pregnant or nursing (lactating) women.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  PFS assessed by BIRC based on RECIST v1.1 .

SECONDARY OUTCOMES:
Overall survival(OS) | Up to 4 years
  OS is defined as the time from the date of randomization to death from any cause.
Objective response rate (ORR) | Up to 2 years
  ORR is the proportion of subjects with CR or PR based on RECIST v1.1.
Duration of response (DoR) | Up to 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1;
Adverse event (AE) | From the time of informed consent signed through 90 days after the last dose of penpulimab
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment
Maximum observed concentration (Cmax) | From first dose of penpulimab through 30 days after last dose of penpulimab
  Serum concentrations of penpulimab in individual subjects at different time points after penpulimab administration.
Anti-drug antibodies (ADA) | From first dose of penpulimab through 30 days after last dose of penpulimab
  Number and percentage of subjects with detectable anti-drug antibody (ADA).
PD-L1 expression | Baseline (Tumor tissue samples must be provided to the research center or central laboratory prior to initial administration).
  Detect PD-L1 expression in tumor samples and evaluate the correlation between PD-L1 and efficacy.
Blood EBV level | Up to 2 years
  Detect the blood EBV level at baseline and changes after administration and evaluate the correlation between EBV and efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Chaosu Hu, MD, Principal Investigator — Fudan University; Xiaozhong Chen, MD, Principal Investigator — Cancer Hospital of The University of Chinese Academy of Sciences
Locations (56):
- United States (5):
  - City of Hope, Duarte, California
  - Winship Cancer Institute/Emory University, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Australia (5):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincent's Public Hospital Sydney, Darlinghurst, New South Wales
  - Genesis Care North Shore, St Leonards, New South Wales
  - Sir Charles Gardner, Heidelberg, Victoria
  - Austin Health, Nedlands, Western Australia
- Brazil (7):
  - Hospital de Câncer de Barretos - Fundação Pio XII, Barretos, REG1
  - Grupo Oncoclínicas, Botafogo, REG1
  - Hospital Bruno Born, Lajeado, REG1
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, REG1
  - Centro de Estudos e Pesquisa de Hematologia, Santo André, REG1
  - Instituto do Câncer do Estado de São Paulo (ICESP), São Paulo, REG1
  - Centro de Câncer A. C. Camargo, São Paulo, REG1
- Canada (2):
  - Alberta Health Services (Tom Baker Cancer Centre), Calgary, Alberta
  - Toronto Sunnybrook Hospital, Toronto, Ontario
- China (37):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Hainan General Hospital, Haikou, Hainan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymized participant data will be considered for sharing once the product and indication have been approved by major health authorities, if there is legal authority to share the data and there is no reasonable likelihood of participant reidentification. Data may be requested from the corresponding author.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol and SAP will be available when the main results of this study are officially published in a scientific journal.
Access Criteria: The study protocol and SAP can be obtained by emailing to the corresponding author of the published paper.